CLINICAL TRIAL: NCT02279823
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Controlled Study to Evaluate the Safety and Efficacy of Cortexolone 17α-Propionate (CB-03-01) Solution 5%, Minoxidil Solution 5%, and Vehicle Solution, Applied Twice-daily for 26 Weeks in Males With Androgenetic Alopecia (AGA)
Brief Title: A Phase 2 Study to Evaluate the Safety and Efficacy of CB-03-01 Solution, a Comparator Solution and Vehicle Solution in Males With Androgenetic Alopecia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Intrepid Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 171-7152-201
Record Dates: First submitted 2014-10-07; First posted 2014-10-31 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Androgenetic Alopecia
Keywords: androgen; alopecia; CB-03-01; solution; topical
MeSH Terms: conditions — Alopecia | interventions — Clascoterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- CB-03-01 solution (Experimental): Topical solution applied twice daily for 26 weeks
  Interventions: Drug: CB-03-01 solution
- Minoxidil Solution 5% (Active Comparator): Topical solution applied twice daily for 26 weeks
  Interventions: Drug: Minoxidil Solution 5%
- Placebo solution (Placebo Comparator): Topical solution applied twice daily for 26 weeks
  Interventions: Drug: Placebo solution

INTERVENTIONS:
Drug: CB-03-01 solution — Investigational drug solution
  Other Names: cortexolone 17α-propionate
  Arms: CB-03-01 solution
Drug: Minoxidil Solution 5% — FDA approved marketed product
  Arms: Minoxidil Solution 5%
Drug: Placebo solution — Vehicle solution
  Arms: Placebo solution

SUMMARY:
In this proof-of-concept study, the safety and efficacy of a solution formulation will be investigated in male subjects with androgenetic alopecia (AGA) after twice daily application for up to 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subject has mild to moderate androgenetic alopecia (AGA) in temple and vertex region
* Subject is willing to maintain the same hairstyle, hair length, and hair color throughout the study
* Subject agrees to continue his other general hair care products and regimen for the entire study
* Subjects who are sexually active with a female partner must be surgically sterile or agree to use an effective method of birth control from the first administration of the test article until 30 days after the last administration

Exclusion Criteria:

* Subject has any dermatological disorders of the scalp in the target region with the possibility of interfering with the application of the test article or examination method, such as fungal or bacterial infections, seborrheic dermatitis, psoriasis, eczema, folliculitis, scars, or scalp atrophy
* Subject has any condition in the opinion of the investigator that could interfere with the evaluation of the test articles or requires the use of interfering topical or systemic therapy (e.g., uncontrolled thyroid disease, certain genetic disorders that involve hair growth or patterns)
* Subject has a current or recent history (within 3 months) of hair transplants, hair weaves or non-breathable wigs and hair bonding
* Subject has a current or recent history (within 3 months) of active hair loss due to diffuse telogen effluvium, alopecia areata, scarring alopecia, trichotillomania or conditions/diseases other than AGA
* Subject has a current or recent history (within 3 months) of severe dietary changes or presenting a history of eating disorder(s)
* Subject has any condition which, in the investigator's opinion, would make it unsafe for the subject to participate in this research study
* Subject is currently enrolled in an investigational drug or device study
* Subject has received an investigational drug or been treated with an investigational device within 30 days prior to the initiation of treatment
* Subject is unable to communicate or cooperate with the investigator due to language problems, poor mental development, or impaired cerebral function
* Subject may be unreliable for the study including subjects who engage in excessive alcohol intake or drug abuse, or subjects who are unable to return for scheduled follow-up visits
* The subject has known hypersensitivity or previous allergic reaction to any of the active or inactive components of the test articles or tattoo ink
* Subject has used any of the following topical preparations or procedures on the scalp:

  * Topical treatments including corticosteroids, pimecrolimus, tacrolimus, minoxidil, hormone therapy, anti-androgens or other agents that are known to affect hair growth in the opinion of the investigator within 12 weeks of the initiation of treatment
  * Topical over-the-counter (OTC) or cosmetic treatments known or reasonably believed to affect hair growth (e.g., brands such as Aminexil, Maxilene, Nioxin, Foltene, etc. or hair health or hair growth products with saw palmetto, copper, etc.) in the opinion of the investigator within 4 weeks of the initiation of treatment.
  * Scalp procedures (surgical, laser, light or energy treatments, etc.) within 6 months of the initiation of treatment
* Subject has used the following systemic medications or procedures:

  * Beta blockers, cimetidine, diazoxide, isotretinoin, vitamin A intake above 10000 IU per day or corticosteroids (including intramuscular and intralesional injections) within 12 weeks of the initiation of treatment. Inhaled, intranasal or ocular corticosteroids are allowed if use is stable (stable use is defined as dose and frequency unchanged for at least 4 weeks prior to the initiation of treatment)
  * Retinoid, cyclosporine therapy within 6 months of the initiation of treatment
  * Finasteride (Propecia®, etc.), dutasteride or a similar product(s) within 12 months of the initiation of treatment
  * Chemotherapy, cytotoxic agents or radiation (of the scalp) within 12 months of the initiation of treatment
  * Other systemic therapy which may materially affect the subject's hair or hair growth in the opinion of the investigator

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2014-10; Primary Completion 2015-12 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change in Target Area Hair Count (TAHC) | Baseline and Month 6
  Changes from Baseline in TAHC [in number of non-vellus hairs] using digital image analysis at Month 6.
Subject Self Assessment (Hair Growth Assessment [HGA]) | Month 6
  The subject's evaluation of treatment benefit via the HGA questionnaires at Month 6. Scalp hair growth is compared from baseline using the following 7-point scale: greatly decreased (-3), moderately decreased (-2), slightly decreased (-1), no change (0), slightly increased (1), moderately increased (2), and greatly increased (3).

SECONDARY OUTCOMES:
Change in Target Area Hair Width (TAHW) | Baseline and Month 6
  Changes from Baseline in TAHW [in μm/cm2] using digital image analysis at Month 6.
Change in Target Area Hair Density (TAHD) | Baseline and Month 6
  Changes from Baseline in TAHD [in intensity units] using digital image analysis at Month 6.
Subject evaluation of treatment benefit via the Hair Growth Index (HGI) and Hair Growth Satisfaction Scale (HGSS) questionnaires | Month 6
  The subject's evaluation of treatment benefit via the HGI and HGSS questionnaires at Month 6.
  HGI: Hair growth is compared from baseline by three questions on a health outcome questionnaire, which are scored using the following 7-point scale: much less (-3), moderately less (-2), slightly less (-1), the same amount (0), slightly more (1), moderately more (2), much more (3).
  HGSS: Hair appearance/growth is compared from baseline by five questions, which are scored using the following 7-point scale: very dissatisfied (-3), dissatisfied (-2), somewhat dissatisfied (-1), neutral/neither satisfied nor dissatisfied (0), somewhat satisfied (1), satisfied (2), very satisfied (3).
Investigator's Global Assessment (IGA) | Baseline, Month 2, 4 and 6
  Compared to Baseline, the investigator will assess the subject's scalp hair growth using the following 7-point scale: greatly decreased (-3), moderately decreased (-2), slightly decreased (-1), no change (0), slightly increased (1), moderately increased (2), and greatly increased (3).

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Andrasfay, Study Director — Therapeutics, Inc.
Locations (3):
- United States (3):
  - Therapeutics Clinical Research, San Diego, California
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - DermResearch, Inc., Austin, Texas